CLINICAL TRIAL: NCT02104843
Title: Effect of Daclatasvir/Asunaprevir/BMS-791325 Three Drug Antiviral Combination Therapy on the Pharmacokinetics of Rosuvastatin
Brief Title: Drug Interaction Between Daclatasvir/Asunaprevir/BMS-791325 and Rosuvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AI443-115
Record Dates: First submitted 2014-04-02; First posted 2014-04-04 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir; asunaprevir; 8-cyclohexyl-N-((dimethylamino)sulfonyl)-1,1a,2,12b-tetrahydro-11-methoxy-1a-((3-methyl-3,8-diazabicyclo(3.2.1)oct-8-yl)carbonyl)cycloprop(d)indolo(2,1-a)(2)benzazepine-5-carboxamide; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1: DCV/ASV/BMS-791325 FDC + BMS-791325 + Rosuvastatin (Experimental): Treatment A: Rosuvastatin tablet orally on specified days
  Treatment B: Daclatasvir, Asunaprevir and BMS-791325 Fixed dose combination (FDC) + BMS-791325 tablet orally on specified days
  Treatment C: Daclatasvir, Asunaprevir and BMS-791325 FDC + BMS-791325 + Rosuvastatin tablet orally on specified days
  Interventions: Drug: Daclatasvir, Asunaprevir and BMS-791325 FDC; Drug: BMS-791325; Drug: Rosuvastatin

INTERVENTIONS:
Drug: Daclatasvir, Asunaprevir and BMS-791325 FDC
Drug: BMS-791325
Drug: Rosuvastatin
  Other Names: Crestor®

SUMMARY:
The primary purpose is to assess the effect of Daclatasvir (DCV)/Asunaprevir (ASV)/BMS-791325 combination therapy on the exposure of Rosuvastatin.

DETAILED DESCRIPTION:
IND Number: 79,599/101,943

Primary Purpose: Other - Phase 1 Clinical Pharmacology drug interaction study in healthy subjects

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy subjects with no clinically significant deviations from normal in medical history, physical exam findings, 12 lead ECG measurements and clinical laboratory tests
* Females must be of non-childbearing potential

Exclusion Criteria:

* Women of childbearing potential
* Any significant acute or chronic medical condition
* Inability to tolerate oral medications
* Inability to be venipunctured and/or tolerate venous access
* Abnormal liver function tests
* Current or recent (within 3 months of dosing) gastrointestinal disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) of Rosuvastatin | Day 1 (predose) to Day 5 (96 hours) and Day 15 (predose) to Day 19 (96 hours)
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (AUC(0-T)) of Rosuvastatin | Day 1 (predose) to Day 5 (96 hours) and Day 15 (predose) to Day 19 (96 hours)
Area under the concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) of Rosuvastatin | Day 1 (predose) to Day 5 (96 hours) and Day 15 (predose) to Day 19 (96 hours)

SECONDARY OUTCOMES:
Time of maximum observed concentration (Tmax) of Rosuvastatin | Days 1 and 15 (predose through 96 hours)
Half life (T-HALF) of Rosuvastatin | Days 1 and 15 (predose through 96 hours)
Apparent total body clearance (CLT/F) of Rosuvastatin | Days 1 and 15 (predose through 96 hours)
Maximum observed concentration (Cmax) of Daclatasvir, Asunaprevir and BMS-791325 and BMS-794712 | Day 15 (predose through 12 hours) and Days 13 and 14 pre-AM-dose
Trough observed plasma concentration (predose) (Ctrough) of Daclatasvir, Asunaprevir and BMS-791325 and BMS-794712 | Day 15 (predose through 12 hours) and Days 13 and 14 pre-AM-dose
Area under the concentration-time curve in one dosing interval [AUC(TAU)] of Daclatasvir, Asunaprevir and BMS-791325 and BMS-794712 | Day 15 (predose through 12 hours) and Days 13 and 14 pre-AM-dose
Time of maximum observed concentration (Tmax) of Daclatasvir, Asunaprevir and BMS-791325 and BMS-794712 | Day 15 (predose through 12 hours) and Days 13 and 14 pre-AM-dose
Observed plasma concentration at 12 hours after dosing in a pharmacokinetic (PK) profile (C12) of Daclatasvir, Asunaprevir and BMS-791325 and BMS-794712 | Day 15 (predose through 12 hours) and Days 13 and 14 pre-AM-dose
Safety measured by incidence of Adverse events (AEs), Serious adverse events (SAEs) and AEs leading to discontinuation | Days 1 through 19
Safety measured by results of vital sign measurements, Electrocardiogram (ECGs), physical examinations and clinical laboratory tests | Days 1 through 19

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb